CLINICAL TRIAL: NCT02503488
Title: Decreasing Youth Involvement in Violence in Burundi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Vivo international e.V. (Industry); Action on Armed Violence (Other); Psychologues sans Frontières Burundi (Other)
Responsible Party: Principal Investigator, Anselm Crombach, Dr. Anselm Crombach, Dipl.-Psych., University of Konstanz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKonstanz
Record Dates: First submitted 2015-06-30; First posted 2015-07-21 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Posttraumatic Stress Disorder; Depression; Aggression
Keywords: Appetitive Aggression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Aggression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Program Group (Experimental): The treatment arm will consist of 20 randomly selected participants who will receive Narrative Exposure Therapy for Forensic Offender Rehabilitation (FORNET) for their traumatic symptomology, aggression, and depression. FORNET consists of a guided exposure of the participant's traumatic experiences in chronological order and integrating them into a coherent biographical memory.The intervention addresses the participant's positive, negative, and violent memories of events that have taken place during their lifetime, and also provides participants an opportunity to asses their current situation and future plans. FORNET can be completed in six sessions and each session lasts 90 minutes on average.
  Interventions: Behavioral: Narrative Exposure Therapy for Forensic Offender Rehab
- Treatment As Usual (TAU) (Active Comparator): Participants in the TAU group will receive group and individual psycho-social support from trained peer-support workers, with 10 sessions occurring throughout the course of the intervention for each participant. In addition, there will be sensitisation trainings as well as mentoring for establishing greater financial independence. Last, TAU will include one-day events promoting social cohesion and peace.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy for Forensic Offender Rehab — See arm description.
  Other Names: FORNET
  Arms: Program Group
Behavioral: Treatment as Usual — See arm description
  Other Names: TAU
  Arms: Treatment As Usual (TAU)

SUMMARY:
The purpose of the current study is to examine the psychological well-being of youth within the context of participation in political violence during the 2015 election period in Burundi. In detail, the investigators are interested in fostering improved outcomes in a peace-building initiative aimed at youth in Burundi by reducing the mental health-related stress of the initiative's most severely affected participants. In addition, the investigators are interested in learning more about the youth experience of involvement in the Burundian political system in an effort to understand the links between youth engagement in political violence and past experiences of traumatic events.

DETAILED DESCRIPTION:
The African Great Lakes Region is marked by several countries which have been ravaged by violence for several years. One of these countries is Burundi, a small state bordered by Rwanda, Tanzania and the Democratic Republic of the Congo. This country has been stricken by more than a decade of civil war, which ended only in 2006.

Today, many people still struggle in coping with the aftermath of the war. Political parties remain largely drawn along ethnic lines. These identities are often manipulated in order to incite violence and intimidation against opposing parties or groups. Violence between rival youth wings was a disturbing feature of the 2010 elections in Burundi, with similar conditions manifesting themselves in advance of the 2015 presidential election.

Further complicating the situation in Burundi, one of the problems people in war-affected populations often face is the high impairment due to mental health problems. Studies in crisis regions have shown that multiple experiences of traumatic life events seriously damages mental health and can lead to disorders such as Posttraumatic Stress Disorder (PTSD) or depression. Further, the risk of developing PTSD rapidly increases with the number of traumatic events experienced, as the occurrence of PTSD is more likely when the accumulation of trauma exceeds a certain limit. This phenomenon has been described as the "building block effect". This means, people in the context of armed conflicts and war are especially at risk to develop PTSD, as the total load of perceived stress is much higher than anywhere else. Furthermore, recent studies have revealed that combatants and other populations living in violent and insecure circumstances may adapt to their environment by developing an attraction to perpetrating violence, i.e. appetitive aggression. While appetitive aggression helps individuals to survive in violent environments by reducing their likelihood of developing trauma-related symptoms, it increases the risk of getting involved in the perpetration of violence.

In order to address the mental health needs of the participants in the present study, the investigators will be utilizing an intervention, Narrative Exposure Therapy for Forensic Offender Rehabilitation (FORNET), that has been demonstrated to reduce posttraumatic symptomology and readiness for aggressive behavior.

Objectives:

The aim of the present study is to investigate the intersection of politics and mental health within the context of Burundi. Specifically, the study will be seeking to answer the following research questions:

1. Mental Health Barriers to Participation in Peace Building Initiatives: What, if any, role does the presence of mental health issues such as PTSD and depression play in effective participation in peace-building efforts? Can FORNET contribute to peace building programs?
2. Links Between Mental Health Issues and Political Participation: What is the role of mental health issues in shaping the readiness to resort to violence as a result of political beliefs and attitudes toward members of other political parties in a post-conflict setting?

   1. Appetitive Aggression. Does the concept of appetitive aggression influence the manner of political participation? Does appetitive aggression have a relationship to the perpetration of politically-motivated violence?
   2. Trauma-related disorders. Do trauma-related disorders such as PTSD and depression influence the manner of political participation? Do they have a relationship to the perpetration of politically-motivated violence?

ELIGIBILITY:
Inclusion Criteria:

* High degree of symptoms of posttraumatic stress disorder according to the Posttraumatic Symptom Scale
* High degree of appetitive aggression
* Violent behavior during the past three months

Exclusion Criteria:

* Current use of mind altering drugs
* Psychotic symptoms

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Baseline PTSD Scores at 3-months-followup and 9-months-followup | Baseline, 3 months, 9 months
  Will be assessed using the PSS-I
Change in Baseline Depression Scores at 3-months-followup and 9-months-followup | Baseline, 3 months, 9 months
  Will be assessed using the Patient Health Questionnaire-9
Change in Baseline Appetitive Aggression Scores at 3-months-followup and 9-months-followup | Baseline, 3 months, 9 months
  Assesses attitudes towards the perception and disposition of different forms of violence using the Appetitive Aggression Scale for Children (AAS-C).

SECONDARY OUTCOMES:
Change in Baseline Physical State at 3-months-followup and 9-months-followup | Baseline, 3 months, 9 months
  Will be assessed using a structured list of a range of ailments
Change in Social Integration Scores at 3-months-followup and 9-months-followup | Baseline, 3 months, 9 months
  Will assess levels of participant integration with family and community using scores between 0-4, with higher scores indicating higher levels of social integration.
Change in Scores on the Attitudes Toward Members of Other Political Parties Scale at 3-months-followup and 9-months-followup | Baseline, 3 months, 9 months
  Will assess nature of attitudes towards other political parties with which the participant is not affiliated.

OTHER OUTCOMES:
Change in Scores on the Opinion on the Civil War Scale at 3-months-followup and 9-months-followup | Baseline, 3 months, 9 months
  Will assess participant opinions on their acceptance of members of other ethnic groups, responsibility for the civil war, and reparation and transitions post-conflict.

CONTACTS AND LOCATIONS:
Overall Officials: Anselm Crombach, Principal Investigator — University of Konstanz, vivo international e.V., Psychologues sans Frontiers Burundi
Locations (1):
- vivo international & Psychologues sans Frontières mental health center, Bujumbura, Burundi